CLINICAL TRIAL: NCT02796365
Title: Prevention Using Exercise Rehabilitation to Offset Cardiac Toxicities Induced Via Chemotherapy
Acronym: HF-PROACTIVE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Collaborators: Helen L. Kay Charitable Trust (Unknown)
Responsible Party: Principal Investigator, Dennis J. Kerrigan, Bioscientific Staff, Henry Ford Health System
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HFHS-HF_PROACTIVE
Record Dates: First submitted 2016-04-29; First posted 2016-06-10 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Doxorubicin Induced Cardiomyopathy; Breast Cancer; Gastric Cancer; Leukemia
Keywords: Exercise; Cancer; Cardiotoxicity; Cardiomyopathy; Cardiac Rehabilitation
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms; Leukemia; Motor Activity; Neoplasms; Cardiotoxicity; Cardiomyopathies | interventions — Exercise

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Exercise (Experimental): Patients will participate in a 10 week outpatient cardiac rehabilitation program. Exercise will consist of 3 days per week of interval training on a treadmill or bike at an intensity between 50-90% of heart rate reserve. Additionally patients will perform resistance exercises 1-2 days per week and attend 8 nutrition and lifestyle classes.
  Interventions: Other: Exercise
- Usual care (No Intervention): Control group will not be instructed on exercise, but encouraged to follow standard medical advice.

INTERVENTIONS:
Other: Exercise — Intervention will include 10 weeks of a standard cardiac rehabilitation program consisting of thrice a week aerobic exercise and 1-2 days per week resistance exercises.
  Arms: Exercise

SUMMARY:
The purpose of this study is to identify patients at risk for future heart failure using novel markers of early cardiac damage and determine if exercise training can improve these emerging markers as well as overall fitness and quality of life.

DETAILED DESCRIPTION:
With more than 14 million cancer survivors in the United States, more patients than ever are living well beyond their initial cancer diagnosis. However despite the tremendous progress, cancer treatments often come with adverse side-effects, perhaps none are more serious or devastating than chemotherapy induced heart failure.

In many patients, the clinical manifestation of heart failure may not appear until a year, or several years, after completion of chemotherapy. While an echocardiogram is part of standardized surveillance for patients on these drugs, current echocardiogram parameters may not be sensitive enough to quickly detect early heart damage which, in some cases, is irreversible.

Unfortunately, even if detected early, there is no uniformity in terms of how to best treat patients with subclinical cardiac dysfunction who are at risk for heart failure. The use of certain blood pressure drugs show promise, especially in patients with hypertension. However, in addition to drug side-effects (e.g. dizziness/lightheadedness), they do not target the underlying mechanism of chemotherapy induced cardiotoxicity.

Exercise, in various forms, has shown promise in animal studies as a potential cardio-protective therapy to counteract drug toxicity. In general, exercise has many pleiotropic effects for patients receiving chemotherapy (e.g. reduces fatigue, improves endurance, reduces frailty, and enhances quality of life). Relative to DOX toxicity, research involving animals has also shown that exercise protects against deleterious heart dysfunction while showing an enhancement of potential mechanisms involved in chemotherapy induced heart failure (i.e. anti-oxidant and anti-apoptosis pathways).

Patients with cancer who receive either doxorubicin (DOX) or trastuzumab will be screened by one of two methods: 1) a strain echo or 2) a high sensitivity troponin. If either test is positive, patients will meet with a board-certified cardiologist who will determine if the patient may participate in the exercise trial. Under the supervision of a trained clinical exercise physiologist patients will undergo baseline testing, which includes: a quality of life assessment via questionaires, a body composition test, cardiopulmonary stress test and a muscle strength test. These assessment will be performed at baseline and at 12 weeks. Also performed at 12 weeks will be a repeat strain echo and high sensitivity troponin.

Following baseline testing patients will be randomized into exercise training versus standard care. The exercise training will include 12 weeks of cardiac rehabilitation which can be offered in Detroit, Livonia, or West Bloomfield. Exercise will consist of 3 days per week of an interval training aerobic exercise on a treadmill and/or bike for 30-60 minutes and 1-2 days per week of an individualized resistance training program.

ELIGIBILITY:
Inclusion Criteria:

* Patients with cancer who are undergoing or have completed the chemotherapy drugs doxorubicin and/or trastuzumab.
* Have had a recent echocardiogram with a relative reduction in LV strain of >10%.
* If no recent echocardiogram, have a troponin value >0.04 ng/mL, or an increase of 0.04 ng/mL if baseline troponin is elevated.
* Age >/= 18 years.
* Eastern Cooperative Oncology Group (ECOG) scale 0-2.
* Males and females.

Exclusion Criteria:

* Patients with an Ejection Fraction <50%
* Patients not deemed appropriate by a cardiologist or oncologist
* Patients with an ECOG scale >2
* Inability to perform exercise
* Patients who already report exercising >2days per week for >29 minutes

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2016-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Left ventricular strain | 12 weeks
  Spectral Doppler measure with General Electric software analysis of global longitudinal strain.

SECONDARY OUTCOMES:
Peak VO2 | 12 weeks
  During a graded treadmill test, breath-by-breath sampling of expired air will be measured using a MGC Diagnostics gas exchange analysis system.
Percent body fat | 12 weeks
  Body fat will be analyzed using air displacement plethysmography (BodPod/Cosmed)
Isokinetic strength | 12 weeks
  Peak torque will be measured using the Biodex Isokinetic dynamometer.
Quality of life | 12 weeks
  Quality of life will be assessed using the Functional Assessment of Cancer Therapy (FACT-G).
Cardiac Troponin | 12 weeks
  High sensitivity cardiac troponin will be analyzed using a commercial immunoassay.

CONTACTS AND LOCATIONS:
Locations (1):
- William Clay Ford Center for Athletic Medicine, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kerrigan DJ, Reddy M, Walker EM, Cook B, McCord J, Loutfi R, Saval MA, Baxter J, Brawner CA, Keteyian SJ. Cardiac Rehabilitation Improves Fitness in Patients With Subclinical Markers of Cardiotoxicity While Receiving Chemotherapy: A RANDOMIZED CONTROLLED STUDY. J Cardiopulm Rehabil Prev. 2023 Mar 1;43(2):129-134. doi: 10.1097/HCR.0000000000000719. Epub 2022 Aug 4. PMID 35940850